CLINICAL TRIAL: NCT03588247
Title: Cerebrovascular EveNts in Patients Undergoing TranscathetER Aortic Valve Implantation With Balloon-expandable Valves Versus Self-expandable Valves.
Acronym: CENTER
Status: Completed | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Jan J. Piek, MD, PhD, Professor, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: CENTER-study
Record Dates: First submitted 2018-07-05; First posted 2018-07-17 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Aortic Valve Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: transcatheter aortic valve implantation — Patients with severe aortic valve stenosis undergo transcatheter aortic valve implantation

SUMMARY:
The aim of this collaborative analysis is to evaluate stroke rates and mortality in patients undergoing TAVI with the self-expandable MCV prosthesis compared to the balloon-expandable ES valve. In the absence of large randomized controlled trials, we will conduct a large collaborative patient-pooled meta-analysis on 30-day stroke and mortality in patients undergoing primary transfemoral TAVI with either MCV or ES valve.

DETAILED DESCRIPTION:
The main aim of this patient-pooled analyses is to compare stroke rates and mortality in patients undergoing TAVI with the self-expandable MCV prosthesis compared to the balloon-expandable ES valve. However, this collaboration may also be used to compare various outcomes.

Studies were included if they complied with the following requirements: original prospective studies, including patients with aortic valve stenosis treated with transfemoral TAVI of native valves and reporting of 30 day stroke outcomes according to VARC criteria or other specified corresponding criteria . Moreover, to be included studies had to report both the use of self-expandable MCV prosthesis and the balloon-expandable ES valve in more than 50 patients in each arm to ensure experience in use of the valves. Studies were excluded if they only addressed patients undergoing valve-in-valve and re-do procedures or bicuspid valves or included the same study population. Principal Investigators of these studies were approached for collaboration.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing transfemoral transcatheter aortic valve procedures

Exclusion Criteria:

* valve-in-valve procedures, other acces routes than transfemoral

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: patients undergoing transfemoral transcatheter aortic valve procedures
Sampling Method: Probability Sample
Enrollment: 12000 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Mortality | 30 days
  Death during the first month after TAVI
Stroke | 30 days
  Stroke during the first month after TAVI

SECONDARY OUTCOMES:
Pacemaker implantation | 30 days
  Pacemaker during the first month after TAVI
Bleeding | 30 days
  Major or life-threatening bleeding during the first month after TAVI
New onset atrial fibrillation | 30 days
  New onset atrial fibrillation during the first month after TAVI
Myocardial infarction | 30 days
  Myocardial infarction during the first month after TAVI

CONTACTS AND LOCATIONS:
Overall Officials: Jan Piek, Prof., Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- Academic Medical Center, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
Collaborators are invited to participate in analyses

REFERENCES:
- [Derived] Aarts HM, van Nieuwkerk AC, Hemelrijk KI, Salgado Fernandez J, Tchetche D, de Brito FS Jr, Barbanti M, Kornowski R, Latib A, D'Onofrio A, Ribichini F, Ferrer MC, Dumonteil N, Abizaid A, Sartori S, D'Errigo P, Tarantini G, Del Sole AP, Orvin K, Pagnesi M, Pinar E, Dangas G, Mehran R, Voskuil M, Delewi R. Surgical Bailout in Patients Undergoing Transfemoral Transcatheter Aortic Valve Replacement: Incidence, Trends, and Clinical Outcomes. JACC Cardiovasc Interv. 2025 Jan 13;18(1):89-99. doi: 10.1016/j.jcin.2024.09.050. PMID 39814498
- [Derived] van Nieuwkerk AC, Aarts HM, Hemelrijk KI, Urbano Carrillo C, Tchetche D, de Brito FS Jr, Barbanti M, Kornowski R, Latib A, D'Onofrio A, Ribichini F, Garcia-Blas S, Dumonteil N, Abizaid A, Sartori S, D'Errigo P, Tarantini G, Lunardi M, Orvin K, Pagnesi M, Navarro F, Dangas G, Mehran R, Delewi R. Cerebrovascular Events in Patients Undergoing Transfemoral Transcatheter Aortic Valve Implantation: A Pooled Patient-Level Study. J Am Heart Assoc. 2024 Sep 3;13(17):e032901. doi: 10.1161/JAHA.123.032901. Epub 2024 Aug 27. PMID 39190595
- [Derived] van Nieuwkerk AC, Aarts HM, Hemelrijk KI, Canton T, Tchetche D, de Brito FS Jr, Barbanti M, Kornowski R, Latib A, D'Onofrio A, Ribichini F, Maneiro Melon N, Dumonteil N, Abizaid A, Sartori S, D'Errigo P, Tarantini G, Fabroni M, Orvin K, Pagnesi M, Vicaino Arellano M, Dangas G, Mehran R, Voskuil M, Delewi R. Bleeding in Patients Undergoing Transfemoral Transcatheter Aortic Valve Replacement: Incidence, Trends, Clinical Outcomes, and Predictors. JACC Cardiovasc Interv. 2023 Dec 25;16(24):2951-2962. doi: 10.1016/j.jcin.2023.10.011. PMID 38151309
- [Derived] van Nieuwkerk AC, Santos RB, Mata RB, Tchetche D, de Brito FS Jr, Barbanti M, Kornowski R, Latib A, D'Onofrio A, Ribichini F, Baan J, Oteo-Dominguez J, Dumonteil N, Abizaid A, Sartori S, D'Errigo P, Tarantini G, Lunardi M, Orvin K, Pagnesi M, Ghattas A, Amat-Santos I, Dangas G, Mehran R, Delewi R. Diabetes mellitus in transfemoral transcatheter aortic valve implantation: a propensity matched analysis. Cardiovasc Diabetol. 2022 Nov 16;21(1):246. doi: 10.1186/s12933-022-01654-x. PMID 36384656
- [Derived] Vlastra W, Jimenez-Quevedo P, Tchetche D, Chandrasekhar J, de Brito FS Jr, Barbanti M, Kornowski R, Latib A, D'Onofrio A, Ribichini F, Baan J, Tijssen JGP, De la Torre Hernandez JM, Dumonteil N, Sarmento-Leite R, Sartori S, Rosato S, Tarantini G, Lunardi M, Orvin K, Pagnesi M, Hernandez-Antolin R, Modine T, Dangas G, Mehran R, Piek JJ, Delewi R. Predictors, Incidence, and Outcomes of Patients Undergoing Transfemoral Transcatheter Aortic Valve Implantation Complicated by Stroke. Circ Cardiovasc Interv. 2019 Mar;12(3):e007546. doi: 10.1161/CIRCINTERVENTIONS.118.007546. PMID 30871358